CLINICAL TRIAL: NCT00634478
Title: Pre-lemniscal Radiation Deep Brain Stimulation for ET
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment. Funding issues.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00008047
Record Dates: First submitted 2008-01-09; First posted 2008-03-13 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Essential Tremor
Keywords: essential tremor; deep brain stimulation
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): preleminiscal radiation deep brain stimulation
  Interventions: Radiation: Pre-lemniscal Radiation Deep Brain Stimulation
- 2 (Active Comparator): VIM deep brain stimulation
  Interventions: Radiation: Pre-lemniscal Radiation Deep Brain Stimulation

INTERVENTIONS:
Radiation: Pre-lemniscal Radiation Deep Brain Stimulation

SUMMARY:
The hypothesis is that prelemniscal radiation (RaPRL) deep brain stimulation (DBS) is more effective for axial (head/neck/voice) tremor, and perhaps, appendicular tremor control in essential tremor patients.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of essential tremor based on clinical criteria established by the Essential Tremor Consortium
2. Moderate or severe axial-dominant (head/neck/voice) tremor (Tremor Rating Scale [TRS] face, tongue, voice, head or trunk tremor score of 2 or above)
3. May have bilateral appendicular tremor
4. Tremor refractory to at least two medications, including primidone and propranolol
5. Age between 21 and 75
6. Male or Female
7. Significant disability due to essential tremor despite medical treatment (TRS score of 2 or above in any one of the items 16-23 [speaking, feeding other than liquids, bringing liquids to mouth, hygiene, dressing, writing, working, and social activities])

Exclusion Criteria:

1. Tremor due to other etiologies
2. Pregnancy
3. Presence of any other neurodegenerative disease
4. Presence of significant cognitive impairment
5. Presence of any medical condition that precludes neurological surgery
6. Patients with another implanted stimulator or metallic implant, e.g. cochlear implant, cardiac pacemaker, spinal cord stimulator, aneurysm clips
7. Patients who have a known need for future MRIs using a full body radio-frequency (RF) coil or a head transmit coil that extends over the chest area or that do not comply with Medtronic's "MRI Guidelines for Medtronic Deep Brain Simulation Systems"
8. Patients with a history of seizures
9. Patients with psychiatric illness that are not well controlled
10. Patients with risk factors for intraoperative or postoperative bleeding (platelet count less than 125,000 per cubic millimeter, PT and PTT not within normal limits)
11. Patients with brain tumors

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01-19 (Actual); Study Completion 2011-01-19 (Actual)

PRIMARY OUTCOMES:
Tremor rating scale axial score and total score | 3 months, 12 months and 24 months

SECONDARY OUTCOMES:
quality of life (SF 36 and clinical global impression of change) | 3 months, 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Serena W Hung, M.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Pahwa R, Lyons KE, Wilkinson SB, Simpson RK Jr, Ondo WG, Tarsy D, Norregaard T, Hubble JP, Smith DA, Hauser RA, Jankovic J. Long-term evaluation of deep brain stimulation of the thalamus. J Neurosurg. 2006 Apr;104(4):506-12. doi: 10.3171/jns.2006.104.4.506. PMID 16619653
- [Background] Putzke JD, Uitti RJ, Obwegeser AA, Wszolek ZK, Wharen RE. Bilateral thalamic deep brain stimulation: midline tremor control. J Neurol Neurosurg Psychiatry. 2005 May;76(5):684-90. doi: 10.1136/jnnp.2004.041434. PMID 15834027
- [Background] Benabid AL, Pollak P, Gao D, Hoffmann D, Limousin P, Gay E, Payen I, Benazzouz A. Chronic electrical stimulation of the ventralis intermedius nucleus of the thalamus as a treatment of movement disorders. J Neurosurg. 1996 Feb;84(2):203-14. doi: 10.3171/jns.1996.84.2.0203. PMID 8592222
- [Background] Kumar R, Lozano AM, Sime E, Lang AE. Long-term follow-up of thalamic deep brain stimulation for essential and parkinsonian tremor. Neurology. 2003 Dec 9;61(11):1601-4. doi: 10.1212/01.wnl.0000096012.07360.1c. PMID 14663050
- [Background] Kitagawa M, Murata J, Uesugi H, Kikuchi S, Saito H, Tashiro K, Sawamura Y. Two-year follow-up of chronic stimulation of the posterior subthalamic white matter for tremor-dominant Parkinson's disease. Neurosurgery. 2005 Feb;56(2):281-9; discussion 281-9. doi: 10.1227/01.neu.0000148167.49105.a3. PMID 15670376
- [Background] Murata J, Kitagawa M, Uesugi H, Saito H, Iwasaki Y, Kikuchi S, Tashiro K, Sawamura Y. Electrical stimulation of the posterior subthalamic area for the treatment of intractable proximal tremor. J Neurosurg. 2003 Oct;99(4):708-15. doi: 10.3171/jns.2003.99.4.0708. PMID 14567607
- [Background] Velasco F, Jimenez F, Perez ML, Carrillo-Ruiz JD, Velasco AL, Ceballos J, Velasco M. Electrical stimulation of the prelemniscal radiation in the treatment of Parkinson's disease: an old target revised with new techniques. Neurosurgery. 2001 Aug;49(2):293-306; discussion 306-8. doi: 10.1097/00006123-200108000-00009. PMID 11504105
- [Background] Plaha P, Patel NK, Gill SS. Stimulation of the subthalamic region for essential tremor. J Neurosurg. 2004 Jul;101(1):48-54. doi: 10.3171/jns.2004.101.1.0048. PMID 15255251